CLINICAL TRIAL: NCT02326935
Title: Proposal for a Non-randomized, Patient Sponsored, Multi-center Study Studying the Impact and Safety of the Utilization of Culture Expanded Autologous, Adipose-derived Mesenchymal Stem Cells Deployed Via Intravenous Injection for the Treatment of Multiple Sclerosis
Brief Title: Multi-Center Study Safety of Adipose Derived Mesenchymal Stem Cells for the Treatment of Multiple Sclerosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: American CryoStem Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRYO-MS-ADSC-006
Record Dates: First submitted 2014-12-18; First posted 2014-12-30 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Multiple Sclerosis
Keywords: MS; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive; Myelitis
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive; Myelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adipose derived mesenchymal cells (Experimental): Intervention: Autologous adipose derived mesenechymal stem cells, 150 million cells deployed via two (2) treatments via intravenous injection
  Other Names:
  ADSC, mesenchymal cells, stromal cells
  Interventions: Biological: Autologous adipose derived mesenchymal cells

INTERVENTIONS:
Biological: Autologous adipose derived mesenchymal cells — Autologous adipose derived mesenchymal cells, 150M cells deployed via two (2) treatments via intravenous injection.
  Other Names: ADSC, mesenchymal cells, stromal cells

SUMMARY:
The intent of this clinical study is to answer the questions: 1) is the proposed treatment safe and 2) is treatment effective in improving the disease pathology of patients with Multiple Sclerosis and clinical outcomes.

DETAILED DESCRIPTION:
This will be an open-label, non-randomized multi-center patient sponsored study of ADSC implantation using an IV delivery system. The study will provide therapies to up to 100 qualified patients who match the inclusion/exclusion criteria, agree to the follow up program and who have provided a signed consent for each procedure.

The treatment is a combination of (a) general detoxification, (b) lymphatic massage/drainage, (c) therapeutic massage, reflexology and acupuncture and (d) cellular infusion therapy in which cells will be deployed via IV injection over two treatments of 60 minutes each during the five (5) day treatment period.

Follow-up data based upon MSIS-29, a modified SF-36 and standard complication questionnaire will be collected at 3, 6 and then annually post treatment by the patients' local physician and reported back to the sponsor where it will be logged into a HIPPA-compliant outcomes database.

Additional safety data, based upon a standard complication questionnaire will be collected via survey of patient at intervals of 3 and 6 months and then annually for a minimum of five (5) years.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Diagnosis of MS
* Aged 18 - 65 years.
* Duration of disease: >5 years
* Signed, written informed consent willing and able to comply with study visits according to protocol for the full study period
* Physically, mentally and legally capable of international travel for treatment

Exclusion Criteria:

* Patients suffering from significant cardiac, renal or hepatic failure or any other disease that may risk the patient or interfere with the ability to interpret the results
* Patient with any active or chronic infection
* No life-threatening organ dysfunction.
* Pregnancy or risk of pregnancy.
* Severe physical limitations or disabilities
* Patients who are seropositive for HIV1, HIV2, Hepatitis B Surface Antigen, and Hepatitis C
* Patients unable to give written informed consent in accordance with research ethics board guidelines
* Treatment with any immunosuppressive therapy within the 3 months prior to randomization
* Current treatment with an investigational therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-11; Primary Completion 2018-05-18 (Actual); Study Completion 2018-05-18 (Actual)

PRIMARY OUTCOMES:
Standard Complication Questionnaire | 3 months
  incidence and nature of adverse events, serious adverse events, or any unanticipated adverse events. The nature, incidence, and rate of adverse events will be assessed
MS Impact Scale - MSIS-29 | 3 months
  Multiple Sclerosis Impact Scale (MSIS-29)
Modified SF-36 Cell-Based Therapy Follow Up | 3 months
  Modified SF-36 for Cell-Based Therapy Follow Up
Physical Evaluation | 3 Months
  Vital signs of sitting blood pressure, temperature and heart rate

SECONDARY OUTCOMES:
MS Impact Scale - MSIS-29 | 6 months
  Multiple Sclerosis Impact Scale (MSIS-29)
MS Impact Scale - MSIS-29 | 1 year
  Multiple Sclerosis Impact Scale (MSIS-29)
Modified SF-36 Cell-Based Therapy Follow Up | 6 months
  Modified SF-36 for Cell-Based Therapy Follow Up
Standard Complication Questionnaire | 6 months
  incidence and nature of adverse events, serious adverse events, or any unanticipated adverse events. The nature, incidence, and rate of adverse events will be assessed
Standard Complication Questionnaire | 1 year
  incidence and nature of adverse events, serious adverse events, or any unanticipated adverse events. The nature, incidence, and rate of adverse events will be assessed
Standard Complication Questionnaire | 2 years
  incidence and nature of adverse events, serious adverse events, or any unanticipated adverse events. The nature, incidence, and rate of adverse events will be assessed
Standard Complication Questionnaire | 3 years
  incidence and nature of adverse events, serious adverse events, or any unanticipated adverse events. The nature, incidence, and rate of adverse events will be assessed
Standard Complication Questionnaire | 4 years
  incidence and nature of adverse events, serious adverse events, or any unanticipated adverse events. The nature, incidence, and rate of adverse events will be assessed
Standard Complication Questionnaire | 5 years
  incidence and nature of adverse events, serious adverse events, or any unanticipated adverse events. The nature, incidence, and rate of adverse events will be assessed
Physical Evaluation | 6 months
  incidence and nature of adverse events, serious adverse events, or any unanticipated adverse events. The nature, incidence, and rate of adverse events will be assessed
Physical Evaluation | 1 Year
  incidence and nature of adverse events, serious adverse events, or any unanticipated adverse events. The nature, incidence, and rate of adverse events will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Louis A Cona, MD, Principal Investigator — The Da Vinci Center
Locations (1):
- The Da Vinci Center, George Town, Cayman Islands